CLINICAL TRIAL: NCT03210961
Title: A PHASE 1, WITHIN COHORT, RANDOMIZED, DOUBLE BLIND, THIRD-PARTY OPEN, PLACEBO-CONTROLLED, SINGLE- AND MULTIPLE DOSE ESCALATION, PARALLEL GROUP STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF PF-06826647 IN HEALTHY SUBJECTS AND SUBJECTS WITH PLAQUE PSORIASIS
Brief Title: A First in Human Study to Evaluate Safety, Tolerability, and Pharmacology of PF-06826647 in Healthy Subjects and Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2501001
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — ropsacitinib; Suspensions

STUDY DESIGN:
Intervention Model Description: Combination single and multiple ascending dose design. Cohorts of participants are assigned to receive interventions based on acceptable safety, tolerability, and pharmacokinetics of previous dose cohort
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-06826647 tablet (Experimental)
  Interventions: Drug: PF-06826647 tablet
- Placebo tablet (Placebo Comparator)
  Interventions: Other: Placebo tablet
- PF-06826647 oral suspension (Experimental)
  Interventions: Drug: PF-06826647 oral suspension
- Placebo oral solution/suspension (Placebo Comparator)
  Interventions: Other: Placebo oral solution/suspension

INTERVENTIONS:
Drug: PF-06826647 tablet — PF-06826647 tablet for oral administration
  Arms: PF-06826647 tablet
Drug: PF-06826647 oral suspension — PF-06826647 suspension for oral administration (oral suspension to be administered to the 3mg starting dose cohort only)
  Arms: PF-06826647 oral suspension
Other: Placebo oral solution/suspension — placebo oral solution for the single ascending dose, first cohort only
  Arms: Placebo oral solution/suspension
Other: Placebo tablet — Matching placebo tablet
  Arms: Placebo tablet

SUMMARY:
This first in human study will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of PF-06826647 in healthy subjects and subjects with plaque psoriasis.

ELIGIBILITY:
Healthy Participants:

Inclusion Criteria:

* Healthy male subjects between ages of 18-55 years
* Healthy female subjects of non-childbearing potential between the ages of 18-55 years
* Body Mass Index (BMI) of 17.5 to 30.5kg/m2; and a total body weight >50kg (110lbs).
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)
* (Optional) Japanese subjects who have four Japanese biologic grandparents born in Japan

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product
* Have a clinically significant infection currently or within 6 months of first dose of study drug

Psoriasis Participants:

Inclusion Criteria:

* Healthy male subjects between ages of 18-65 years
* Healthy female subjects of non-childbearing potential between the ages of 18-65 years
* Have a diagnosis of plaque psoriasis for at least 6 months prior to first study dose
* Have plaque-type psoriasis covering at least 15% of total body surface area (BSA) at Day-1(prior to randomization in the study
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)

Exclusion Criteria:

* Currently have non-plaque forms of psoriasis, eg, erythrodermic, guttate, or pustular psoriasis
* Have a clinically significant infection currently or within 6 months of first dose of study drug, or a history of chronic or recurrent infectious disease
* Pregnant female subjects; breastfeeding female subjects; female subjects of childbearing potential
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Tehlirian C, Peeva E, Kieras E, Scaramozza M, Roberts ES, Singh RSP, Pradhan V, Banerjee A, Garcet S, Xi L, Gale JD, Vincent MS, Krueger J. Safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of the oral TYK2 inhibitor PF-06826647 in participants with plaque psoriasis: a phase 1, randomised, double-blind, placebo-controlled, parallel-group study. Lancet Rheumatol. 2021 Mar;3(3):e204-e213. doi: 10.1016/S2665-9913(20)30397-0. Epub 2020 Dec 24. PMID 38279383
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2501001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 208 potential participants were screened after signing an informed consent form, of whom 109 participants were randomized to receive study treatment.
Groups:
- Placebo (PBO) SAD (3 Milligrams [mg], 10 mg): During the SAD period (Period 1), healthy participants received placebo matching PF-06826647 3, or 10 mg single dose (SD) cohort in fasted state.
- PBO SAD Followed by (->) PBO QD MAD: During SAD period (Period 1), healthy participants received placebo matching PF-06826647 30, 100, 400, or 1600 mg SD cohort, respectively, in fasted state. At least 14 days separated the beginning of the SAD and MAD periods. In MAD period (Period 2), these participants received placebo matching PF-06826647 30, 100, 400, or 1600 mg once daily (QD) cohort, respectively, for 10 days with standard meal.
- PBO QD MAD Japanese Cohort (JP): During the MAD period (Period 2), Japanese healthy participants received placebo matching PF-06826647 400 mg QD MAD JP cohort with standard meal. MAD period duration was 28 days.
- PBO Twice Daily (BID): During the MAD period (Period 2), healthy participants received placebo matching PF-06826647 200 mg BID cohort with standard meal.
- PF-06826647 3 mg SAD: During the SAD period (Period 1), healthy participants received PF-06826647 3 mg SD in fasted state. SAD period duration was 8 days.
- PF-06826647 10 mg SAD: During the SAD period (Period 1), healthy participants received PF-06826647 10 mg SD in fasted state. SAD period duration was 8 days.
- PF-06826647 30 mg SAD -> 30 mg QD MAD: During the SAD period (Period 1), healthy participants received PF-06826647 30 mg SD in fasted state. At least 14 days separated the beginning of the SAD and MAD periods. In the MAD period (Period 2), these healthy participants received PF-06826647 30 mg QD for 10 days with standard meal. SAD period duration was 8 days and MAD period duration was 28 days.
- PF-06826647 100 mg SAD -> 100 mg QD MAD: During the SAD period (Period 1), healthy participants received PF-06826647 100 mg SD in fasted state. At least 14 days separated the beginning of the SAD and MAD periods. In the MAD period (Period 2), these healthy participants 4 received PF-06826647 100 mg QD for 10 days with standard meal. SAD period duration was 8 days and MAD period duration was 28 days.
- PF-06826647 400 mg SAD -> 400 mg QD MAD: During the SAD period (Period 1), healthy participants received PF-06826647 400 mg SD in fasted state. At least 14 days separated the beginning of the SAD and MAD periods. In the MAD period (Period 2), these healthy participants received PF-06826647 400 mg QD for 10 days with standard meal. SAD period duration was 8 days and MAD period duration was 28 days. SAD period duration was 8 days and MAD period duration was 28 days.
- PF-06826647 1600 mg SAD -> 1200 mg QD MAD: During the SAD period (Period 1), healthy participants received PF-06826647 1600 mg SD in fasted state. At least 14 days separated the beginning of the SAD and MAD periods. In the MAD period (Period 2), these healthy participants received PF-06826647 1200 mg QD for 10 days with standard meal. SAD period duration was 8 days and MAD period duration was 28 days.
- PF-06826647 200 mg BID: During the MAD period (Period 2), healthy participants received PF-06826647 200 mg BID for 10 days with standard meal. MAD period duration was 28 days.
- PF-06826647 400 mg QD MAD JP: During the MAD period (Period 2), Japanese healthy participants received PF-06826647 400 mg QD for 10 days with standard meal. MAD period duration was 28 days.
- PBO QD Psoriasis Cohort (PSO): In the psoriasis placebo cohorts, psoriasis participants received placebo matching PF-06826647 400, or 100 mg QD cohort, respectively, for 28 days with standard meal. Psoriasis cohorts duration was 84 days, safety and AE evaluations lasted up to Day 84, while vital signs, physical, and laboratory abnormality evaluations lasted up to Day 56.
- PF-06826647 400 mg QD PSO: In this psoriasis cohort, psoriasis participants received PF-06826647 400 mg QD for 28 days with standard meal. Psoriasis cohorts duration was 84 days, safety and AE evaluations lasted up to Day 84, while vital signs, physical, and laboratory abnormality evaluations lasted up to Day 56.
- PF-06826647 100 mg QD PSO: In this psoriasis cohort, psoriasis participants received PF-06826647 100 mg QD for 28 days with standard meal. Psoriasis cohorts duration was 84 days, safety and AE evaluations lasted up to Day 84, while vital signs, physical, and laboratory abnormality evaluations lasted up to Day 56.
Period: Overall Study
Arm/Group | Placebo (PBO) SAD (3 Milligrams [mg], 10 mg) | PBO SAD Followed by (->) PBO QD MAD | PBO QD MAD Japanese Cohort (JP) | PBO Twice Daily (BID) | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD -> 30 mg QD MAD | PF-06826647 100 mg SAD -> 100 mg QD MAD | PF-06826647 400 mg SAD -> 400 mg QD MAD | PF-06826647 1600 mg SAD -> 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP | PBO QD Psoriasis Cohort (PSO) | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO
Started | 4 | 9 | 1 | 2 | 6 | 6 | 8 | 7 | 8 | 6 | 7 | 5 | 14 | 15 | 11
Completed | 4 | 9 | 1 | 1 | 6 | 6 | 7 | 7 | 8 | 6 | 6 | 5 | 12 | 11 | 9
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study medication.
Groups:
- Placebo (PBO) SAD (3 mg, 10 mg): During the SAD period (Period 1), healthy participants received placebo matching PF-06826647 3, or 10 mg single dose (SD) cohort in fasted state.
- PBO BID: During the MAD period (Period 2), healthy participants received placebo matching PF-06826647 200 mg BID cohort with standard meal.
- Total: Total of all reporting groups
Arm/Group | Placebo (PBO) SAD (3 mg, 10 mg) | PBO SAD Followed by (->) PBO QD MAD | PBO QD MAD Japanese Cohort (JP) | PBO BID | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD -> 30 mg QD MAD | PF-06826647 100 mg SAD -> 100 mg QD MAD | PF-06826647 400 mg SAD -> 400 mg QD MAD | PF-06826647 1600 mg SAD -> 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP | PBO QD Psoriasis Cohort (PSO) | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO | Total
Number analyzed (Participants) | 4 | 9 | 1 | 2 | 6 | 6 | 8 | 7 | 8 | 6 | 7 | 5 | 14 | 15 | 11 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (12.23) | 42.2 (10.84) | 34.0 (NA) — only 1 participant in this cohort | 32.5 (4.95) | 44.3 (11.47) | 40.2 (10.30) | 40.5 (11.64) | 36.9 (7.40) | 37.5 (8.23) | 31.2 (5.00) | 37.4 (9.27) | 39.8 (5.40) | 38.3 (13.25) | 40.9 (11.62) | 39.0 (13.39) | 39.0 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Male | 4 | 8 | 1 | 2 | 6 | 5 | 8 | 7 | 7 | 6 | 7 | 5 | 14 | 15 | 11 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 4 | 2 | 0 | 7 | 4 | 8 | 40
  Not Hispanic or Latino | 2 | 4 | 1 | 2 | 6 | 6 | 5 | 6 | 4 | 2 | 5 | 5 | 7 | 11 | 3 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 5 | 1 | 3 | 0 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 3 | 0 | 0 | 2 | 4 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 17
  White | 3 | 6 | 0 | 1 | 3 | 1 | 6 | 3 | 6 | 5 | 4 | 0 | 11 | 9 | 11 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vital Signs Data Meeting Pre-Specified Criteria (Single Ascending Dose [SAD] Period)
Description: Maximum absolute values and changes from baseline for vital signs (for supine systolic/diastolic blood pressure [BP] and supine pulse rate [PR]) were summarized descriptively by treatment. Numbers of participants meeting the categorical criteria were provided.
  Number of participants in PBO SAD cohorts = number of participants in [PBO SAD (3mg, 10mg)] cohorts + number of participants in [PBO SAD -> PBO QD MAD] cohorts.
Time Frame: Baseline up to Day 8
Population: The analysis population included the healthy participants who received study treatment and who had the safety parameters in the SAD Period. MAD and Psoriasis Cohorts data were not included.
Measure: Count of Participants; unit: Participants
Groups:
- PBO SAD: During the SAD period (Period 1), healthy participants received placebo matching PF-06826647 3, 10, 30, 100, 400, or 1600 mg single dose (SD) cohort in fasted state. Participants in PBO SAD cohorts = participants in [PBO SAD (3mg, 10mg)] cohorts + participants in [PBO SAD -> PBO QD] cohorts.
- PF-06826647 3 mg SAD: During the SAD period (Period 1), healthy participants received PF-06826647 3 mg SD in fasted state.
- PF-06826647 10 mg SAD: During the SAD period (Period 1), healthy participants received PF-06826647 10 mg SD in fasted state.
- PF-06826647 30 mg SAD: During the SAD period (Period 1), healthy participants received PF-06826647 30 mg SD in fasted state.
- PF-06826647 100 mg SAD: During the SAD period (Period 1), healthy participants received PF-06826647 100 mg SD in fasted state.
- PF-06826647 400 mg SAD: During the SAD period (Period 1), healthy participants received PF-06826647 400 mg SD in fasted state.
- PF-06826647 1600 mg SAD: During the SAD period (Period 1), healthy participants received PF-06826647 1600 mg SD in fasted state.
Arm/Group | PBO SAD | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 13 | 6 | 6 | 8 | 7 | 8 | 6
Participants
  Supine diastolic BP Value <50 mmHg | 2 | 2 | 1 | 0 | 1 | 0 | 0
  Supine diastolic BP Change (Chg) ≥20 mmHg increase | 3 | 1 | 1 | 2 | 1 | 0 | 2
  Supine diastolic BP Chg ≥20 mmHg decrease | 2 | 1 | 2 | 1 | 2 | 1 | 0
  Supine pulse rate Value <40 beats per minute (bpm) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Supine pulse rate Value >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine systolic BP Value <90mmHg | 1 | 1 | 2 | 1 | 0 | 0 | 0
  Supine systolic BP Chg ≥30 mmHg increase | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Supine systolic BP Chg ≥30mmHg decrease | 2 | 1 | 1 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Vital Signs Data Meeting Pre-Specified Criteria (Multiple Ascending Dose [MAD] Period)
Description: Maximum absolute values and changes from baseline for vital signs (for supine systolic/diastolic blood pressure and supine pulse rate) were summarized descriptively by treatment. Numbers of participants meeting the categorical criteria were provided.
Time Frame: Baseline up to Day 28
Population: The analysis population included the healthy participants who received study treatment in the MAD Period. The PBO QD MAD sequence is comprised of both non-Japanese and Japanese participants. The non-Japanese participants had completed the SAD period and continued into the MAD period. The Japanese participants took part only in the MAD period.
Measure: Count of Participants; unit: Participants
Groups:
- PBO QD MAD (JP PBO Included): This arm includes both non-Japanese and Japanese participants. In MAD period (Period 2), the non-Japanese participants received placebo matching PF-06826647 30, 100, 400, or 1200 mg once daily (QD) cohort while the Japanese participants received placebo matching PF-06826647 400 mg QD Japanese cohort, both for 10 days with standard meal.
- PF-06826647 30 mg QD MAD: In the MAD period (Period 2), these healthy participants received PF-06826647 30 mg QD for 10 days with standard meal.
- PF-06826647 100 mg QD MAD: In the MAD period (Period 2), these healthy participants received PF-06826647 100 mg QD for 10 days with standard meal.
- PF-06826647 400 mg QD MAD: In the MAD period (Period 2), these healthy participants received PF-06826647 400 mg QD for 10 days with standard meal.
- PF-06826647 1200 mg QD MAD: In the MAD period (Period 2), these healthy participants received PF-06826647 1200 mg QD for 10 days with standard meal.
Arm/Group | PBO QD MAD (JP PBO Included) | PBO BID | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 400 mg QD MAD | PF-06826647 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP
Number analyzed (Participants) | 9 | 2 | 6 | 6 | 6 | 5 | 7 | 5
Participants
  Supine diastolic BP Value < 50 mmHg | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Supine diastolic BP Chg ≥ 20 mmHg increase | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 0
  Supine diastolic BP Chg ≥ 20 mmHg decrease | 4 | 0 | 2 | 1 | 1 | 1 | 1 | 2
  Supine pulse rate Value < 40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine pulse rate Value > 120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine systolic blood pressure Value < 90 mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Supine systolic BP Chg ≥ 30 mmHg increase | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0
  Supine systolic BP Chg ≥ 30 mmHg decrease | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Vital Signs Data Meeting Pre-Specified Criteria (Psoriasis Cohorts)
Description: as for outcome 2
Time Frame: Baseline up to Day 56
Population: The analysis population included the psoriasis participants who received study treatment and who had the safety parameters in the Psoriasis Cohorts. Data in SAD/MAD Periods were not included.
Measure: Count of Participants; unit: Participants
Groups:
- PBO QD PSO: In the psoriasis (PSO) cohorts, psoriasis participants received placebo matching PF-06826647 400, or 100 mg QD PSO cohort for 28 days with standard meal.
- PF-06826647 400 mg QD PSO: In this psoriasis cohort, psoriasis participants received PF-06826647 400 mg QD for 28 days with standard meal. Psoriasis cohort duration was 84 days.
- PF-06826647 100 mg QD PSO: In this psoriasis cohort, psoriasis participants received PF-06826647 100 mg QD for 28 days with standard meal. Psoriasis cohort duration was 84 days.
Arm/Group | PBO QD PSO | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO
Number analyzed (Participants) | 14 | 15 | 11
Participants
  Supine diastolic blood pressure Value < 50 mmHg | 0 | 1 | 1
  Supine diastolic BP Chg ≥ 20 mmHg increase | 0 | 3 | 5
  Supine diastolic BP Chg ≥ 20 mmHg decrease | 6 | 7 | 4
  Supine pulse rate Value < 40 bpm | 0 | 0 | 0
  Supine pulse rate Value > 120 bpm | 0 | 0 | 0
  Supine systolic BP Value < 90 mmHg | 1 | 0 | 0
  Supine systolic BP Chg ≥ 30 mmHg increase | 0 | 1 | 2
  Supine systolic BP Chg ≥ 30 mmHg decrease | 6 | 5 | 1

4. Primary Outcome: Number of Participants With Physical Examination Data Meeting Pre-Specified Criteria (SAD Period)
Description: Physical examinations were conducted by a physician, trained physician assistant, or nurse practitioner as acceptable according to local regulation. A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The examination assessed the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. Findings were considered to be clinically significant based on investigator's decision.
  Number of participants in PBO SAD cohorts = number of participants in [PBO SAD (3mg, 10mg)] cohorts + number of participants in [PBO SAD -> PBO QD MAD] cohorts.
Time Frame: Baseline up to Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PBO SAD | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 13 | 6 | 6 | 8 | 7 | 8 | 6
Participants
  cardiovascular | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ears | 0 | 0 | 0 | 0 | 0 | 0 | 0
  eyes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  gastrointestinal | 0 | 0 | 0 | 0 | 0 | 0 | 0
  general appearance | 0 | 0 | 0 | 0 | 0 | 0 | 0
  head | 0 | 0 | 0 | 0 | 0 | 0 | 0
  heart | 0 | 0 | 0 | 0 | 0 | 0 | 0
  lungs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  lymph nodes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  mouth | 0 | 0 | 0 | 0 | 0 | 0 | 0
  musculoskeletal | 0 | 0 | 0 | 0 | 0 | 0 | 0
  neurological | 0 | 0 | 0 | 0 | 0 | 0 | 0
  nose | 0 | 0 | 0 | 0 | 0 | 0 | 0
  skin | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Physical Examination Data Meeting Pre-Specified Criteria (MAD Period)
Description: Physical examinations were conducted by a physician, trained physician assistant, or nurse practitioner as acceptable according to local regulation. A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The examination assessed the participants for any potential changes in general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. Findings were considered to be clinically significant based on investigator's decision.
Time Frame: Baseline up to Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- PBO QD MAD: This arm includes both non-Japanese and Japanese participants. In MAD period (Period 2), the non-Japanese participants received placebo matching PF-06826647 30, 100, 400, or 1200 mg once daily (QD) cohort while the Japanese participants received placebo matching PF-06826647 400 mg QD Japanese cohort, both for 10 days with standard meal.
Arm/Group | PBO QD MAD | PBO BID | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 400 mg QD MAD | PF-06826647 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP
Number analyzed (Participants) | 9 | 2 | 6 | 6 | 6 | 5 | 7 | 5
Participants
  cardiovascular | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ears | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  eyes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  gastrointestinal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  general appearance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  head | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  heart | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  lungs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  lymph nodes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  mouth | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  musculoskeletal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  neurological | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  nose | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  skin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Physical Examination Data Meeting Pre-Specified Criteria (Psoriasis Cohorts)
Description: as for outcome 5
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PBO QD PSO | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO
Number analyzed (Participants) | 14 | 15 | 11
Participants
  cardiovascular | 0 | 0 | 0
  ears at screening | 0 | 0 | 0
  ears at Day 28 | 0 | 1 | 0
  eyes | 0 | 0 | 0
  gastrointestinal | 0 | 0 | 0
  general appearance | 0 | 0 | 0
  head | 0 | 0 | 0
  heart | 0 | 0 | 0
  lungs | 0 | 0 | 0
  lymph nodes | 0 | 0 | 0
  mouth | 0 | 0 | 0
  musculoskeletal | 0 | 0 | 0
  neurological | 0 | 0 | 0
  nose | 0 | 0 | 0
  skin | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-Specified Criteria (SAD Period)
Description: ECG endpoints and changes from baseline (QTcF, PR and QRS) were summarized descriptively by cohort and treatment using pre-defined categories. Numbers of participants meeting the categorical criteria were provided. All planned and unplanned post-dose time points were counted in these categorical summaries. Categorical summarization criteria for ECG were as follows: 1) QTcF maximum absolute value ≥450 and <480 millisecond (msec), ≥480 and <500 msec. ≥500 msec; 2) QTcF maximum increase ≥30 and <60 msec, ≥60 msec; 3) PR maximum absolute value ≥300 msec; 4) PR maximum increases from baseline ≥25% if baseline >200 msec, ≥50% if baseline ≤200 msec; 5) QRS maximum absolute value ≥140 msec; 6) QRS maximum increase from baseline ≥50%.
  Number of participants in PBO SAD cohorts = number of participants in [PBO SAD (3mg, 10mg)] cohorts + number of participants in [PBO SAD -> PBO QD MAD] cohorts.
Time Frame: Baseline up to Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PBO SAD | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 13 | 6 | 6 | 8 | 7 | 8 | 6
Participants
  PR maximum absolute value ≥300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR maximum increase from baseline ≥25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS maximum absolute value ≥140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS maximum increase from baseline ≥50% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF maximum absolute value ≥450 and <480 msec | 0 | 0 | 0 | 0 | 0 | 1 | 0
  QTCF maximum absolute value ≥480 and <500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF maximum absolute value ≥500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF maximum increase ≥30 and <60 msec | 0 | 1 | 0 | 0 | 1 | 0 | 0
  QTCF maximum increase from baseline ≥60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With ECG Data Meeting Pre-Specified Criteria (MAD Period)
Description: ECG endpoints and changes from baseline (QTcF, PR and QRS) were summarized descriptively by cohort and treatment using pre-defined categories. Numbers of participants meeting the categorical criteria were provided. All planned and unplanned post-dose time points were counted in these categorical summaries. Categorical summarization criteria for ECG were as follows: 1) QTcF maximum absolute value ≥450 and <480 millisecond (msec), ≥480 and <500 msec. ≥500 msec; 2) QTcF maximum increase ≥30 and <60 msec, ≥60 msec; 3) PR maximum absolute value ≥300 msec; 4) PR maximum increases from baseline ≥25% if baseline >200 msec, ≥50% if baseline ≤200 msec; 5) QRS maximum absolute value ≥140 msec; 6) QRS maximum increase from baseline ≥50%.
Time Frame: Baseline up to Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PBO QD MAD | PBO BID | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 400 mg QD MAD | PF-06826647 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP
Number analyzed (Participants) | 9 | 2 | 6 | 6 | 6 | 5 | 7 | 5
Participants
  PR maximum absolute value ≥300 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR maximum increase from baseline ≥25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS maximum absolute value ≥140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS maximum increase from baseline ≥50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF maximum absolute value ≥450 and <480 msec | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  QTCF maximum absolute value ≥480 and <500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF maximum absolute value ≥500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF maximum increase ≥30 and <60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF maximum increase from baseline ≥60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With ECG Data Meeting Pre-Specified Criteria (Psoriasis Cohorts)
Description: as for outcome 8
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PBO QD PSO | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO
Number analyzed (Participants) | 14 | 15 | 11
Participants
  PR maximum absolute value ≥300 msec | 0 | 0 | 0
  PR maximum increase from baseline ≥25/50% | 0 | 0 | 0
  QRS maximum absolute value ≥140 msec | 0 | 0 | 0
  QRS maximum increase from baseline ≥50% | 0 | 0 | 0
  QTCF maximum absolute value ≥450 and <480 msec | 0 | 0 | 0
  QTCF maximum absolute value ≥480 and <500 msec | 0 | 0 | 0
  QTCF maximum absolute value ≥500 msec | 0 | 0 | 0
  QTCF maximum increase ≥30 and <60 msec | 0 | 0 | 0
  QTCF maximum increase from baseline ≥60 msec | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Who Withdrew Due to Adverse Events (AEs) (SAD Period)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. All events occurring following start of the treatment or increasing in severity were counted as treatment emergent. Events that occurred in a non-treatment period (eg, washout or follow-up) were counted as treatment emergent and attributed to the previous treatment taken. For each event, the investigator pursued and obtained adequate information both to determine the outcome and to assess whether it meets the criteria for classification as an SAE.
  PBO SAD cohorts = [PBO SAD (3mg, 10mg)] cohorts + [PBO SAD -> PBO QD MAD] cohorts.
Time Frame: Baseline up to Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PBO SAD | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 13 | 6 | 6 | 8 | 7 | 8 | 6
Participants
  Participants with AEs (AC) | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Participants with AEs (TR) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Participants with SAEs (AC) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with SAEs (TR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with severe AEs (AC) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with severe AEs (TR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants withdrew due to AEs (AC) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants withdrew due to AEs (TR) | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With TEAEs, SAEs, and Who Withdrew Due to AEs (MAD Period)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening (immediate risk of death); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. All events occurring following start of the treatment or increasing in severity were counted as treatment emergent. Events that occurred in a non-treatment period (eg, washout or follow-up) were counted as treatment emergent and attributed to the previous treatment taken. For each event, the investigator pursued and obtained adequate information both to determine the outcome and to assess whether it meets the criteria for classification as an SAE.
Time Frame: Baseline up to Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PBO QD MAD | PBO BID | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 400 mg QD MAD | PF-06826647 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP
Number analyzed (Participants) | 9 | 2 | 6 | 6 | 6 | 5 | 7 | 5
Participants
  Participants with AEs (AC) | 2 | 0 | 2 | 1 | 1 | 1 | 3 | 1
  Participants with AEs (TR) | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1
  Participants with SAEs (AC) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with SAEs (TR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with severe AEs (AC) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with severe AEs (TR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants withdrew due to AEs (AC) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participants withdrew due to AEs (TR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With TEAEs, SAEs, and Who Withdrew Due to AEs (Psoriasis Cohorts)
Description: as for outcome 11
Time Frame: Baseline up to Day 84
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PBO QD PSO | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO
Number analyzed (Participants) | 14 | 15 | 11
Participants
  Participants with AEs (AC) | 7 | 12 | 5
  Participants with AEs (TR) | 5 | 5 | 3
  Participants with SAEs (AC) | 0 | 0 | 0
  Participants with SAEs (TR) | 0 | 0 | 0
  Participants with severe AEs (AC) | 0 | 0 | 0
  Participants with severe AEs (TR) | 0 | 0 | 0
  Participants withdrew due to AEs (AC) | 0 | 1 | 0
  Participants withdrew due to AEs (TR) | 0 | 1 | 0

13. Primary Outcome: Number of Participants With Laboratory Abnormalities (SAD Period)
Description: Laboratory data were listed and summarized by treatment in accordance with the sponsor reporting standards. Parameters for laboratory abnormalities evaluation included: erythrocyte mean corpuscular volume (Ery. MCV), erythrocyte mean corpuscular hemoglobin (Ery. MCH), reticulocytes/erythrocytes (%), limphocytes, eosinophils, bilirubin, aspartate aminotransferase (AST), urate, high-density lipoproteins (HDL) cholesterol, low-density lipoproteins (LDL) cholesterol, triglycerides, cholesterol, ketones, nitrite, leukocyte esterase, epithelial cells, urinalysis-bacteria.
  Number of participants in PBO SAD cohorts = number of participants in [PBO SAD (3mg, 10mg)] cohorts + number of participants in [PBO SAD -> PBO QD MAD] cohorts.
Time Frame: Baseline up to Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PBO SAD | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 13 | 6 | 6 | 8 | 7 | 8 | 6
Participants
  Ery. MCV (femtoliters [fL]) <0.9 × LLN | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Ery. MCH (picograms [pg]) <0.9 × LLN | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Reticulocytes/erythrocytes (%) >1.5 x ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Limphocytes (10^3/mm^3) <0.8 × LLN | 0 | 0 | 1 | 0 | 1 | 1 | 0
  Eosinophils (10^3/mm^3) >1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bilirubin (mg/dL) >1.5 x ULN | 0 | 0 | 0 | 1 | 0 | 0 | 0
  AST (U/L) >3 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urate (mg/dL) >1.2 x ULN | 0 | 0 | 1 | 0 | 0 | 0 | 0
  HDL cholesterol (mg/dL) <0.8 × LLN | 0 | 0 | 0 | 0 | 0 | 1 | 0
  LDL cholesterol (mg/dL) >1.2 x ULN | 10 | 4 | 3 | 6 | 2 | 5 | 4
  Triglycerides (mg/dL) >1.3 x ULN | 2 | 2 | 1 | 2 | 1 | 2 | 2
  Cholesterol (mg/dL) >1.3 x ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Ketones ≥1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Nitrite ≥1 | 2 | 0 | 0 | 0 | 0 | 2 | 1
  Leukocyte esterase ≥1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Epithelial cells (/LPF) ≥6: number analyzed (Participants) | 2 | 1 | 1 | 0 | 0 | 2 | 2
  Epithelial cells (/LPF) ≥6 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Urinalysis-bacteria (/HPF) ≥20: number analyzed (Participants) | 2 | 1 | 1 | 0 | 0 | 2 | 2
  Urinalysis-bacteria (/HPF) ≥20 | 1 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Laboratory Abnormalities (MAD Period)
Description: Laboratory data were listed and summarized by treatment in accordance with the sponsor reporting standards. Parameters and corresponding primary criteria for laboratory abnormalities evaluation included: Ery. MCV <0.9 × LLN, Ery. Mean corpuscular hemoglobin (Ery. MCH) <0.9 × LLN or >1.1 ULN, reticulocytes/erythrocytes (%) >1.5 × ULN, lymphocytes <0.8 × LLN or >1.2 × ULN, neutrophils <0.8 × LLN, eosinophils >1.2 × ULN, bilirubin >1.5 × ULN, urate >1.2 × ULN, HDL cholesterol <0.8 × LLN, LDL cholesterol >1.2 × ULN, triglycerides >1.3 × ULN, bicarbonate >1.1 × ULN, cholesterol >1.3 × ULN, urine glucose ≥1, urine hemoglobin ≥1, nitrite ≥1, leukocyte esterase ≥1, epithelial cells ≥6/LPF, urinalysis-casts >1/LPF, urinalysis-bacteria >20/HPF, urine 24 hours creatinine >1.1 × ULN.
Time Frame: Baseline up to Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PBO QD MAD | PBO BID | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 400 mg QD MAD | PF-06826647 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP
Number analyzed (Participants) | 9 | 2 | 6 | 6 | 6 | 5 | 7 | 5
Participants
  Ery. MCV (fL) <0.9 × LLN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Ery. MCH (pg) <0.9 × LLN | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Ery. MCH (pg) >1.1 × ULN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Reticulocytes/erythrocytes (%) >1.5 × ULN | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocytes (10^3/mm^3) <0.8 × LLN | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Lymphocytes (10^3/mm^3) >1.2 × ULN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils (10^3/mm^3) <0.8 × LLN | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
  Eosinophils (10^3/mm^3) >1.2 x ULN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Bilirubin (mg/dL) >1.5 x ULN | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Urate (mg/dL) >1.2 x ULN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  HDL cholesterol (mg/dL) <0.8 × LLN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  LDL cholesterol (mg/dL) >1.2 x ULN | 7 | 1 | 4 | 2 | 5 | 4 | 5 | 5
  Triglycerides (mg/dL) >1.3 x ULN | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 2
  Bicarbonate (mEq/L) >1.1 x ULN | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
  cholesterol (mg/dL) >1.3 x ULN | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
  Urine glucose ≥1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Urine hemoglobin ≥1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Nitrite ≥1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
  Leukocyte esterase ≥1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Epithelial cells (/LPF) ≥6: number analyzed (Participants) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1
  Epithelial cells (/LPF) ≥6 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urinalysis-casts (/LPF) >1: number analyzed (Participants) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1
  Urinalysis-casts (/LPF) >1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urinalysis-bacteria (/HPF) >20: number analyzed (Participants) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1
  Urinalysis-bacteria (/HPF) >20 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urine 24 hours creatinine (mg/24 hr) >1.1 x ULN: number analyzed (Participants) | 9 | 1 | 5 | 6 | 6 | 5 | 6 | 5
  Urine 24 hours creatinine (mg/24 hr) >1.1 x ULN | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With Laboratory Abnormalities (Psoriasis Cohorts)
Description: Laboratory data were listed and summarized by treatment in accordance with the sponsor reporting standards. Parameters and corresponding primary criteria for laboratory abnormalities evaluation included: reticulocytes/erythrocytes (%) >1.5 × ULN, lymphocytes <0.8 × LLN, neutrophils <0.8 × LLN or >1.2 × ULN, eosinophils >1.2 × ULN, bilirubin >1.5 × ULN, alanine aminotransferase (ALT) >3.0 × ULN, creatinine >1.3 × ULN, urate >1.2 × ULN, HDL cholesterol <0.8 × LLN, LDL cholesterol >1.2 × ULN, triglycerides >1.3 × ULN, potassium >1.1 × ULN, bicarbonate >1.1 × ULN, glucose <0.6 × LLN or >1.5 × ULN, Creatine Kinase (CK) >2.0 × ULN, cholesterol >1.3 × ULN, urine glucose ≥1, ketones ≥1, urine hemoglobin ≥1, urine bilirubin ≥1, leukocyte esterase ≥1, epithelial cells ≥6/LPF, urinalysis-bacteria/HPF.
Time Frame: Baseline up to Day 56
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PBO QD PSO | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO
Number analyzed (Participants) | 14 | 15 | 11
Participants
  Reticulocytes/erythrocytes (%) >1.5 x ULN | 2 | 3 | 1
  Lymphocytes (10^3/mm^3) <0.8 x LLN | 1 | 1 | 0
  Neutrophils (10^3/mm^3) <0.8 x LLN | 0 | 1 | 0
  Neutrophils (10^3/mm^3) >1.2 x ULN | 1 | 0 | 1
  Eosinophils (10^3/mm^3) >1.2 x ULN | 1 | 1 | 1
  Bilirubin (mg/dL) >1.5 x ULN | 0 | 1 | 0
  ALT (U/L) >3 x ULN | 0 | 0 | 1
  Creatinine (mg/dL) >1.3 x ULN | 0 | 0 | 1
  Urate (mg/dL) >1.2 x ULN | 7 | 6 | 3
  HDL cholesterol (mg/dL) <0.8 x LLN | 0 | 1 | 0
  LDL cholesterol (mg/dL) >1.2 x ULN | 11 | 8 | 6
  Triglycerides (mg/dL) >1.3 x ULN | 6 | 4 | 3
  Potassium (mEq/L) >1.1 x ULN | 0 | 0 | 1
  Bicarbonate (mEq/L) >1.1 x ULN | 2 | 0 | 0
  Glucose (mg/dL) <0.6 x LLN | 1 | 0 | 0
  Glucose (mg/dL) >1.5 x ULN | 1 | 0 | 0
  CK (U/L) >2 x ULN | 4 | 2 | 3
  cholesterol (mg/dL) >1.3 x ULN | 0 | 1 | 1
  Urine glucose ≥1 | 0 | 0 | 1
  Ketones ≥1 | 1 | 1 | 0
  Urine hemoglobin ≥1 | 0 | 1 | 2
  Urine bilirubin ≥1 | 0 | 0 | 1
  Leukocyte esterase ≥1 | 2 | 0 | 1
  Epithelial cells (/LPF) ≥6: number analyzed (Participants) | 4 | 1 | 3
  Epithelial cells (/LPF) ≥6 | 3 | 0 | 0
  Urinalysis-bacteria (/HPF) >20: number analyzed (Participants) | 4 | 1 | 3
  Urinalysis-bacteria (/HPF) >20 | 0 | 0 | 1

16. Primary Outcome: Change in 24 Hour Creatinine Clearance From Day -1 on Day 10 (MAD Period)
Description: Change in 24-hour creatinine clearance at Day 10 from Day -1 (baseline) during the MAD was presented by treatment group.
Time Frame: Day -1 and Day 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliters per minute (mL/min)
Arm/Group | PBO QD MAD | PBO BID | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 400 mg QD MAD | PF-06826647 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP
Number analyzed (Participants) | 9 | 1 | 5 | 6 | 6 | 5 | 6 | 5
milliliters per minute (mL/min) | -21.0 (98.76) | -32.0 (NA) — One (1) participant was analyzed, so standard deviation did not exist. | -62.4 (45.10) | 0.2 (65.64) | -52.5 (56.22) | -11.4 (58.76) | -64.7 (36.22) | 40.2 (45.26)

17. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) (SAD Period)
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time 0 (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: The analysis population included the healthy participants who received study treatment and who had the PK parameter in the SAD Period. MAD and Psoriasis Cohorts data were not included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per mL (ng*hr/mL)
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 7 | 4
nanograms*hours per mL (ng*hr/mL) | 47.63 (59) | 369.3 (67) | 848.4 (40) | 1582 (42) | 3056 (65) | 11790 (25)

18. Secondary Outcome: Secondary: Dose Normalized AUCinf (AUCinf[dn]) (SAD Period)
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time 0 (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf). AUCinf(dn) = AUCinf / dose. Dose normalized AUC values of PF-06826647 was plotted against dose and included individual participant values and the geometric means for each dose. These plots were used to help understand the relationship between the plasma PK parameters and dose.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 7 | 4
ng*hr/mL/mg | 15.86 (59) | 36.93 (67) | 28.28 (41) | 15.82 (42) | 7.636 (65) | 7.370 (25)

19. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to 24 Hours (AUC24) (SAD Period)
Description: AUC24 was summarized by dosing regimen and period. It was determined by linear/log trapezoidal method.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 8 | 6
ng*hr/mL | 43.10 (56) | 347.8 (62) | 543.2 (49) | 1158 (55) | 2519 (67) | 9318 (34)

20. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) (SAD Period)
Description: AUClast was summarized by dosing regimen and period. It was determined by linear/log trapezoidal method.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 8 | 6
ng*hr/mL | 40.25 (56) | 354.8 (67) | 638.5 (58) | 1375 (53) | 2767 (65) | 9921 (32)

21. Secondary Outcome: Dose Normalized AUClast (AUClast[dn]) (SAD Period)
Description: AUClast(dn) = AUClast / dose. Dose normalized AUC values of PF-06826647 were plotted against dose and included individual participant values and the geometric means for each dose. These plots was used to help understand the relationship between the plasma PK parameters and dose.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 8 | 6
ng*hr/mL/mg | 13.40 (56) | 35.48 (67) | 21.28 (58) | 13.75 (53) | 6.919 (65) | 6.200 (32)

22. Secondary Outcome: Maximum Plasma Concentration (Cmax) (SAD Period)
Description: Cmax was summarized by dosing regimen and period. It was observed directly from data.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 8 | 6
ng/mL | 7.844 (38) | 47.09 (35) | 77.93 (34) | 166.8 (55) | 404.8 (62) | 1218 (25)

23. Secondary Outcome: Dose Normalized Cmax (Cmax[dn]) (SAD Period)
Description: Cmax(dn) = Cmax / dose. To assess the relationship between Cmax and dose, dose normalized Cmax was plotted against dose, and included individual participant values and the geometric means for each dose.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: The analysis population included healthy participants who received the study treatment and who had the PK parameter in the SAD Period. MAD and Psoriasis Cohorts data were not included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 8 | 6
ng/mL/mg | 2.617 (38) | 4.709 (35) | 2.597 (34) | 1.668 (55) | 1.012 (62) | 0.7618 (25)

24. Secondary Outcome: Time for Cmax (Tmax) (SAD Period)
Description: Tmax was summarized by dosing regimen and period. It was observed directly from data as time of first occurrence.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 23
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 8 | 6
hours (hr) | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [2.00 to 6.00] | 2.00 [0.500 to 4.00] | 2.00 [0.500 to 4.00]

25. Secondary Outcome: Terminal Elimination Half-Life ((t½) (SAD Period)
Description: t1/2 was summarized by dosing regimen and period. It was determined by loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve. Only those data points judged to describe the terminal log linear decline were used in the regression.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 7 | 4
hours (hr) | 3.620 (1.2956) | 6.032 (1.9050) | 19.69 (9.5144) | 38.77 (35.966) | 16.25 (9.3430) | 22.21 (24.586)

26. Secondary Outcome: Mean Residence Time (MRT) (SAD Period)
Description: MRT = AUMCinf / AUCinf, where AUMCinf is the area under the first moment curve from time 0 to infinity.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (hr)
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 7 | 4
hours (hr) | 5.596 (26) | 7.761 (30) | 16.97 (43) | 21.23 (81) | 10.56 (36) | 9.417 (33)

27. Secondary Outcome: Apparent Volume of Distribution (Vz/F) (SAD Period)
Description: Vz/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 7 | 4
liters (L) | 312.1 (34) | 226.1 (41) | 902.9 (81) | 2671 (134) | 2732 (128) | 2877 (146)

28. Secondary Outcome: Apparent Clearance (CL/F) (SAD Period)
Description: CL/F is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24,36,48,72,168 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Arm/Group | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 100 mg SAD | PF-06826647 400 mg SAD | PF-06826647 1600 mg SAD
Number analyzed (Participants) | 5 | 6 | 6 | 3 | 7 | 4
liters per hour (L/hr) | 62.98 (59) | 27.08 (67) | 35.36 (41) | 63.21 (42) | 130.8 (65) | 135.4 (26)

29. Secondary Outcome: Area Under the Plasma Concentration-Time Profile Over the Dosing Interval τ (AUCτ) (MAD Period Day 1)
Description: AUCτ was summarized by dosing regimen and period. Dosing interval was the interval τ between administration of doses of drug. In this study, the dosing interval was 24 hours for QD dosing and 12 hours for BID dosing. It was determined by linear/log trapezoidal method.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: The analysis population included healthy participants who received study treatment on Day 1 and who had the Day 1 PK parameters in the MAD Period. Data on the other days of MAD Period as well as in SAD and Psoriasis Cohorts were not included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- PF-06826647 200 mg BID MAD: During the MAD period (Period 2), healthy participants received PF-06826647 200 mg BID for 10 days with standard meal.
- PF-06826647 400 QD MAD: In the MAD period (Period 2), these healthy participants in Cohort 5 received PF-06826647 400 mg QD for 10 days with standard meal.
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 5 | 5
ng*hr/mL | 662.8 (25) | 1803 (23) | 1646 (70) | 4424 (67) | 6038 (29) | 17090 (20)

30. Secondary Outcome: Dose Normalized AUCτ (AUCτ[dn]) (MAD Period Day 1)
Description: Area Under the Plasma Concentration-Time Profile over the Dosing interval τ (AUCτ). Dosing interval was the interval τ between administration of doses of drug. In this study, the dosing interval τ was 24 hours for QD dosing and 12 hours for BID dosing.
  AUCτ(dn) = AUCτ / Dose. To assess the relationship between the PK parameters and the dose, dose normalized AUCτ was plotted against dose, and included individual participant values and the geometric means for each dose.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 5 | 5
ng*hr/mL/mg | 22.10 (25) | 18.03 (23) | 8.229 (70) | 11.07 (67) | 15.10 (29) | 14.23 (20)

31. Secondary Outcome: Cmax (MAD Period Day 1)
Description: Cmax was summarized by dosing regimen and period. It was observed directly from data.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 5 | 5
ng/mL | 83.53 (24) | 267.2 (20) | 289.8 (67) | 585.9 (33) | 695.5 (19) | 2023 (10)

32. Secondary Outcome: Cmax(dn) (MAD Period Day 1)
Description: as for outcome 23
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 5 | 5
ng/mL/mg | 2.787 (24) | 2.672 (20) | 1.450 (67) | 1.468 (33) | 1.741 (19) | 1.686 (10)

33. Secondary Outcome: Tmax (MAD Period Day 1)
Description: Tmax was summarized by dosing regimen and period. It was observed directly from data as time of first occurrence.
Time Frame: Day 1 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 29
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 5 | 5
hours (hr) | 3.00 [2.00 to 6.00] | 4.00 [1.00 to 4.00] | 4.00 [2.00 to 6.00] | 3.00 [2.00 to 6.00] | 4.00 [2.00 to 4.00] | 2.00 [2.00 to 4.00]

34. Secondary Outcome: AUCτ (MAD Period Day 10)
Description: as for outcome 29
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: The analysis population included healthy participants who received study treatment on Day 10 and who had the Day 10 PK parameters in the MAD Period. Data on the other days of MAD Period as well as in SAD and Psoriasis Cohorts were not included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ng*hr/mL | 752.9 (32) | 1952 (33) | 2010 (49) | 5420 (57) | 7194 (20) | 14890 (31)

35. Secondary Outcome: AUCτ(dn) (MAD Period Day 10)
Description: as for outcome 30
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ng*hr/mL/mg | 25.06 (32) | 19.52 (33) | 10.04 (49) | 13.56 (57) | 18.00 (19) | 12.41 (31)

36. Secondary Outcome: Cmax (MAD Period Day 10)
Description: Cmax was summarized by dosing regimen and period. It was observed directly from data.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ng/mL | 85.34 (27) | 263.2 (30) | 339.5 (46) | 667.3 (37) | 887.0 (11) | 1855 (21)

37. Secondary Outcome: Cmax(dn) (MAD Period Day 10)
Description: as for outcome 23
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ng/mL/mg | 2.844 (27) | 2.632 (30) | 1.701 (46) | 1.669 (37) | 2.220 (11) | 1.547 (21)

38. Secondary Outcome: Tmax (MAD Period Day 10)
Description: Tmax was summarized by dosing regimen and period. It was observed directly from data as time of first occurrence.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
hours (hr) | 4.00 [4.00 to 6.00] | 4.00 [2.00 to 4.00] | 4.00 [2.00 to 4.00] | 4.00 [2.00 to 6.00] | 4.00 [2.00 to 6.00] | 4.00 [2.00 to 4.00]

39. Secondary Outcome: Average Concentration at Steady State (Cav) (MAD Period Day 10)
Description: Cav = AUCτ,ss / τ, where ss means 'at steady state', and where the dosing interval τ was 24 hours for QD dosing and 12 hours for BID dosing. Cav was summarized by dosing regimen and period.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ng/mL | 31.36 (32) | 81.28 (34) | 167.6 (49) | 226.0 (57) | 299.7 (20) | 619.9 (31)

40. Secondary Outcome: Lowest Concentration Observed During the Dosing Interval τ (Cmin) (MAD Period Day 10)
Description: Cmin was observed directly from data. It was summarized by dosing regimen and period. Dosing interval was the interval τ between administration of doses of drug. In this study, the dosing interval τ was 24 hours for QD dosing and 12 hours for BID dosing.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ng/mL | 6.273 (83) | 10.40 (75) | 55.01 (65) | 24.77 (148) | 29.50 (60) | 62.26 (112)

41. Secondary Outcome: Terminal Elimination Half-Life ((t½) (MAD Period Day 10)
Description: as for outcome 25
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24,48,72,96,168 hours post-dose
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 5 | 3 | 4 | 4 | 5
hours (hr) | 8.802 (5.8142) | 12.72 (12.644) | 26.93 (8.1132) | 7.500 (2.5803) | 7.433 (4.7975) | 34.33 (21.926)

42. Secondary Outcome: MRT (MAD Period Day 10)
Description: MRT = AUMCinf / AUCinf, where AUMCinf is the area under the first moment curve from time 0 to infinity.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24,48,72,96,168 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (hr)
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 5 | 3 | 4 | 4 | 5
hours (hr) | 10.56 (44) | 9.872 (33) | 17.14 (26) | 9.622 (26) | 7.996 (19) | 9.165 (24)

43. Secondary Outcome: Peak Trough Ratio (PTR) (MAD Period Day 10)
Description: PTR = Cmax,ss / Cmin,ss, where ss means 'at steady state'. It was summarized by dosing regimen and period.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ratio | 13.61 (69) | 25.31 (55) | 6.951 (23) | 26.92 (112) | 30.09 (61) | 29.76 (97)

44. Secondary Outcome: Observed Accumulation Ratio Based on AUC (Rac) (MAD Period Day 10)
Description: Rac = AUCτ,ss / AUCτ,sd, where ss means 'at steady state' and sd 'single dose'. In this study, Rac = AUCτ(Day 10) / AUCτ(Day 1). Rac was summarized by dosing regimen and period.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ratio | 1.085 (8) | 1.082 (21) | 1.328 (52) | 1.225 (39) | 1.191 (24) | 0.8711 (30)

45. Secondary Outcome: Observed Accumulation Ratio Based on Cmax (Rac,Cmax) (MAD Period Day 10)
Description: Rac,Cmax = Cmax,ss / Cmax,sd, where ss means 'at steady state' and sd 'single dose'. In this study, Rac,Cmax = Cmax(Day10) / Cmax(Day 1). Rac,Cmax was summarized by dosing regimen and period.
Time Frame: Days 1 and 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
ratio | 0.9295 (22) | 0.9852 (24) | 1.282 (57) | 1.139 (35) | 1.275 (14) | 0.9176 (25)

46. Secondary Outcome: Vz/F (MAD Period Day 10)
Description: as for outcome 27
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 5 | 3 | 4 | 4 | 5
liters (L) | 433.5 (52) | 643.6 (98) | 3224 (90) | 758.9 (93) | 519.2 (67) | 2944 (166)

47. Secondary Outcome: CL/F (MAD Period Day 10)
Description: as for outcome 28
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
liters per hour (L/hr) | 39.86 (32) | 51.27 (34) | 99.47 (49) | 73.78 (57) | 55.62 (20) | 80.63 (31)

48. Secondary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine From Time 0 to the Dosing Interval τ Hours Post-Dose (Aeτ) (MAD Period Day 10)
Description: Dosing interval was the interval τ between administration of doses of drug. In this study, the dosing interval τ was 24 hours for QD dosing and 12 hours for BID dosing. Aeτ = Sum of [urine concentration * sample volume] for each collection interval. Aer was summarized by dosing regimen and period.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
mg | 0.2204 (35) | 1.072 (65) | 2.560 (66) | 3.134 (75) | 2.931 (624) | 14.73 (92)

49. Secondary Outcome: Percentage of Dose Recovered Unchanged in Urine From Time 0 to the Dosing Interval τ Hours Post-Dose (Aeτ%) (MAD Period Day 10)
Description: Dosing interval was the interval τ between administration of doses of drug. In this study, the dosing interval τ was 24 hours for QD dosing and 12 hours for BID dosing. Aeτ% = Aeτ / Dose * 100. Aeτ%was summarized by dosing regimen and period.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Dose
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
Percentage of Dose | 0.7344 (35) | 1.072 (65) | 1.280 (66) | 0.7827 (75) | 0.7333 (624) | 1.228 (92)

50. Secondary Outcome: Renal Clearance (Clr) (MAD Period Day 10)
Description: Renal clearance was calculated as cumulative amount of drug recovered unchanged in urine during the dosing interval (Aeτ) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCτ), where dosing interval is 24 hours for QD dosing and 12 hours for BID dosing.
Time Frame: Day 10 pre-dose, and 0.5,1,2,4,6,8,12,24 hours post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06826647 30 mg QD MAD | PF-06826647 100 mg QD MAD | PF-06826647 200 mg BID MAD | PF-06826647 400 QD MAD | PF-06826647 400 mg QD MAD JP | PF-06826647 1200 mg QD MAD
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 5 | 5
L/hr | 0.2928 (70) | 0.5500 (42) | 1.274 (39) | 0.5777 (34) | 0.4076 (500) | 0.9909 (58)

51. Secondary Outcome: AUCτ (Psoriasis Cohorts)
Description: AUCτ was summarized by dosing regimen and period. It was determined by linear/log trapezoidal method.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: The analysis population included psoriasis participants who received study treatment on Day 1 and who had the Day 1 PK parameters in the Psoriasis Cohorts. Data on the other days of Psoriasis Cohorts study treatment period, as well as in SAD/MAD Periods were not included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
ng*hr/mL | 2401 (53) | 7664 (34)

52. Secondary Outcome: AUCτ(dn) (Psoriasis Cohorts)
Description: AUCτ(dn) = AUCτ / Dose. To assess the relationship between the PK parameters and the dose, dose normalized AUCτ was plotted against dose, and included individual participant values and the geometric means for each dose.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
ng*hr/mL/mg | 24.01 (53) | 19.17 (34)

53. Secondary Outcome: Cmax (Psoriasis Cohorts)
Description: Cmax was summarized by dosing regimen and period. It was observed directly from data.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
ng/mL | 296.6 (38) | 869.8 (25)

54. Secondary Outcome: Cmax(dn) (Psoriasis Cohorts)
Description: Cmax was summarized by dosing regimen and period. It was observed directly from data.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
ng/mL/mg | 2.966 (38) | 2.176 (25)

55. Secondary Outcome: Tmax (Psoriasis Cohorts)
Description: Tmax was summarized by dosing regimen and period. It was observed directly from data as time of first occurrence.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
hours (hr) | 4.00 [1.00 to 6.00] | 4.00 [2.00 to 6.00]

56. Secondary Outcome: Cav (Psoriasis Cohorts)
Description: Cav = AUCτ,ss / τ, where ss means 'at steady state'. Cav was summarized by dosing regimen and period.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
ng/mL | 100.2 (53) | 319.3 (34)

57. Secondary Outcome: Cmin (Psoriasis Cohorts)
Description: Cmin was observed directly from data. It was summarized by dosing regimen and period.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
ng/mL | 21.92 (103) | 38.12 (176)

58. Secondary Outcome: Terminal Elimination Half-Life ((t½) (Psoriasis Cohorts)
Description: as for outcome 25
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24,168 hours post-dose
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 11
hours (hr) | 7.796 (5.7087) | 6.809 (5.4050)

59. Secondary Outcome: MRT (Psoriasis Cohorts)
Description: MRT = AUMCinf / AUCinf, where AUMCinf is the area under the first moment curve from time 0 to infinity.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24,168 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (hr)
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 11
hours (hr) | 11.27 (41) | 9.444 (28)

60. Secondary Outcome: PTR (Psoriasis Cohorts)
Description: PTR = Cmax,ss / Cmin,ss, it was summarized by dosing regimen and period.
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
ratio | 13.52 (76) | 22.81 (171)

61. Secondary Outcome: Vz/F (Psoriasis Cohorts)
Description: as for outcome 27
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 11
liters (L) | 408.1 (30) | 461.2 (54)

62. Secondary Outcome: CL/F (Psoriasis Cohorts)
Description: as for outcome 28
Time Frame: Day 28 pre-dose, and 0.5,1,2,4,6,8,12,16,24 hours post-dose
Population: as for outcome 51
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06826647 100 mg QD PSO | PF-06826647 400 mg QD PSO
Number analyzed (Participants) | 10 | 13
L/hr | 41.61 (53) | 52.21 (34)

63. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Day 28
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections: head, arms, trunk, legs. For each section, percent area of skin involved was estimated: 0= 0% to 6= 90-100%. Severity was estimated by clinical signs: erythema, induration, desquamation; scale: 0= none to 4= maximum. Final PASI = sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0= no disease to 72= maximal disease.
Time Frame: Baseline and Day 28
Population: The analysis population included psoriasis participants who received the 28-day study treatment and who had the efficacy parameters at Baseline and on Day 28 in the Psoriasis Cohorts. Data in SAD/MAD Periods were not included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PBO QD PSO | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO
Number analyzed (Participants) | 12 | 13 | 11
score on a scale | -11.13 (2.405) | -24.18 (2.281) | -14.62 (2.505)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 8 for SAD Cohorts, which included PF-06826647 3mg, 10mg, 30mg, 100mg, 400mg, and 1600mg SD cohorts as well as placebo matching each SAD cohort. Baseline up to Day 28 for MAD Cohorts, which included PF-06826647 30mg, 100mg, 400mg, 1200mg QD, 200mg BID, 400mg QD JP, as well as placebo matching each MAD cohort. Baseline up to Day 84 for Psoriasis Cohorts, which included PF-06826647 400mg and 100mg QD cohorts, as well as placebo matching each psoriasis cohort.
Description: The requirements for recording safety events on the CRF and for reporting safety events on the Clinical Trial Serious Adverse Event Report Form to Pfizer Safety were delineated for 3 types of events: (1) SAEs; (2) non-serious adverse events (AEs); and (3) exposure to the investigational product under study during pregnancy or breastfeeding, and occupational exposure.
Groups:
- Placebo SAD: During the SAD period (Period 1), the healthy participants received placebo matching PF-06826647 3, 10, 30, 100, 400, or 1600 mg cohort SD cohort in fasted state. SAD period duration was 8 days. (Those placebo participants matching 30, 100, 400, or 1600 SD cohort later continued into MAD period and received the placebo matching 30, 100, 400, or 1200 mg QD cohort, respectively.)
- Placebo QD MAD (JP Placebo Included): This arm includes both non-Japanese and Japanese participants. In MAD period (Period 2), the non-Japanese participants (they had completed the SAD period) received placebo matching PF-06826647 30, 100, 400, or 1200 mg QD cohort while the Japanese participants (they did not take part in SAD period) received placebo matching PF-06826647 400 mg QD Japanese cohort, both for 10 days with standard meal. MAD period duration was 28 days.
- Placebo BID: Edit During the MAD period (Period 2), the healthy participants received placebo matching PF-06826647 200 mg BID cohort for 10 days with standard meal. MAD period duration was 28 days.
- PF-06826647 3 mg SAD: During the SAD period (Period 1), the healthy participants received PF-06826647 3 mg SD in fasted state. SAD period duration was 8 days.
- PF-06826647 10 mg SAD: During the SAD period (Period 1), the healthy participants received PF-06826647 10 mg SD in fasted state. SAD period duration was 8 days.
- PF-06826647 30 mg SAD: During the SAD period (Period 1), the healthy participants received PF-06826647 30 mg SD in fasted state. SAD period duration was 8 days. (These participants later continued into PF-06826647 30 mg QD in MAD period.)
- PF-06826647 30 mg QD MAD: During the MAD period (Period 2), the healthy participants who had taken PF-06826647 30 mg SD received PF-06826647 30 mg QD for 10 days with standard meal. MAD period duration was 28 days.
- PF-06826647 100 mg SAD: During the SAD period (Period 1), the healthy participants received PF-06826647 100 mg SD in fasted state. SAD period duration was 8 days. (These participants later continued into PF-06826647 100 mg QD in MAD period.)
- PF-06826647 100 mg QD MAD: During the MAD period (Period 2), the healthy participants who had taken PF-06826647 100 mg SD received PF-06826647 100 mg QD for 10 days with standard meal. MAD period duration was 28 days.
- PF-06826647 400 mg SAD: During the SAD period (Period 1), the healthy participants received PF-06826647 400 mg SD in fasted state. SAD period duration was 8 days. (These participants later continued into PF-06826647 400 mg QD in MAD period.)
- PF-06826647 400 mg QD MAD: During the MAD period (Period 2), the healthy participants who had taken PF-06826647 400 mg SD received PF-06826647 400 mg QD for 10 days with standard meal. MAD period duration was 28 days.
- PF-06826647 1600 mg SAD: During the SAD period (Period 1), the healthy participants received PF-06826647 1600 mg SD in fasted state. SAD period duration was 8 days. (These participants later continued into PF-06826647 1200 mg QD in MAD period.)
- PF-06826647 1200 mg QD MAD: During the MAD period (Period 2), the healthy participants who had taken PF-06826647 1600 mg SD received PF-06826647 1200 mg QD for 10 days with standard meal. MAD period duration was 28 days.
- PF-06826647 200 mg BID: During the MAD period (Period 2), the healthy participants received PF-06826647 200 mg BID for 10 days with standard meal. MAD period duration was 28 days.
- PF-06826647 400 mg QD MAD JP: During the MAD period (Period 2), the Japanese healthy participants received PF-06826647 400 mg QD for 10 days with standard meal. MAD period duration was 28 days.
- Placebo QD PSO: In the psoriasis (PSO) cohorts, the psoriasis participants received placebo matching PF-06826647 400, or 100 mg QD PSO cohort for 28 days with standard meal. Psoriasis cohort duration was 84 days.
- PF-06826647 400 mg QD PSO: In this psoriasis cohort, the psoriasis participants received PF-06826647 400 mg QD for 28 days with standard meal. Psoriasis cohort duration was 84 days.
- PF-06826647 100 mg QD PSO: In this psoriasis cohort, the psoriasis participants received PF-06826647 100 mg QD for 28 days with standard meal. Psoriasis cohort duration was 84 days.
Arm/Group | Placebo SAD | Placebo QD MAD (JP Placebo Included) | Placebo BID | PF-06826647 3 mg SAD | PF-06826647 10 mg SAD | PF-06826647 30 mg SAD | PF-06826647 30 mg QD MAD | PF-06826647 100 mg SAD | PF-06826647 100 mg QD MAD | PF-06826647 400 mg SAD | PF-06826647 400 mg QD MAD | PF-06826647 1600 mg SAD | PF-06826647 1200 mg QD MAD | PF-06826647 200 mg BID | PF-06826647 400 mg QD MAD JP | Placebo QD PSO | PF-06826647 400 mg QD PSO | PF-06826647 100 mg QD PSO
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9 | 0/2 | 0/6 | 0/6 | 0/8 | 0/6 | 0/7 | 0/6 | 0/8 | 0/6 | 0/6 | 0/5 | 0/7 | 0/5 | 0/14 | 0/15 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9 | 0/2 | 0/6 | 0/6 | 0/8 | 0/6 | 0/7 | 0/6 | 0/8 | 0/6 | 0/6 | 0/5 | 0/7 | 0/5 | 0/14 | 0/15 | 0/11
Other Adverse Events (participants affected / at risk) | 1/13 | 2/9 | 0/2 | 0/6 | 0/6 | 0/8 | 2/6 | 1/7 | 1/6 | 0/8 | 1/6 | 2/6 | 1/5 | 3/7 | 1/5 | 7/14 | 12/15 | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SAD (N=13) | Placebo QD MAD (JP Placebo Included) (N=9) | Placebo BID (N=2) | PF-06826647 3 mg SAD (N=6) | PF-06826647 10 mg SAD (N=6) | PF-06826647 30 mg SAD (N=8) | PF-06826647 30 mg QD MAD (N=6) | PF-06826647 100 mg SAD (N=7) | PF-06826647 100 mg QD MAD (N=6) | PF-06826647 400 mg SAD (N=8) | PF-06826647 400 mg QD MAD (N=6) | PF-06826647 1600 mg SAD (N=6) | PF-06826647 1200 mg QD MAD (N=5) | PF-06826647 200 mg BID (N=7) | PF-06826647 400 mg QD MAD JP (N=5) | Placebo QD PSO (N=14) | PF-06826647 400 mg QD PSO (N=15) | PF-06826647 100 mg QD PSO (N=11)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 3 (5) | 2 (2)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03210961/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT03210961/SAP_001.pdf